CLINICAL TRIAL: NCT06004011
Title: Integrated Delivery of Cancer Control Interventions for Adolescents and Young Adults Living With HIV in Zambia
Brief Title: AYAHIV Role-based Responsibilities for Oncology-focused Workforce (ARROW)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Implenomics (Other)
Collaborators: Population Council (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Imp001
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer; Kaposi Sarcoma; Non Hodgkin Lymphoma
Keywords: cancer screening; Implementation trial
MeSH Terms: conditions — Uterine Cervical Neoplasms; Sarcoma, Kaposi; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARROW strategies (Experimental): The ARROW strategies which use peer-peer support at the patient level (through peer counselors), at the provider level (through peer lead education sessions) and at the health system level (through a health collaborative forum) to deliver high quality screenings and ensure cancer treatment completion.
  Interventions: Other: ARROW strategies
- One-time education (Active Comparator): The comparator arm participants will receive one-time education and usual care services.
  Interventions: Other: One-time education

INTERVENTIONS:
Other: ARROW strategies — ARROW strategies are peer-to-peer support at the patient, provider and health system levels
  Arms: ARROW strategies
Other: One-time education — The comparison group will receive a one-time education campaign that will provide informational brochures to adolescents and young adults living with HIV and HIV providers
  Arms: One-time education

SUMMARY:
Adolescents and young adults living with HIV experience higher premature mortality from cancer than their uninfected peers. In Zambia, because of multilevel barriers, interventions for early diagnosis and optimized treatment to reduce this cancer mortality are underutilized for this disproportionally impacted cohort. In this study, the investigators will test peer-to-peer education and support strategies to increase use of early diagnosis services in HIV treatment facilities and improve compliance with cancer treatment in the cancer center.

DETAILED DESCRIPTION:
Zambia is a global epicenter for HIV with a large number of adolescents and young adults living with HIV (AYAHIV). Compared with their uninfected peers, AYAHIV are at increased risk of developing cancer, most frequently Kaposi sarcoma (KS), non-Hodgkin's lymphoma (NHL), and cervical cancer (CC). To reduce this premature mortality, evidence-based strategies should be implemented to both diagnose cancers at an earlier stage and help AYAHIV complete recommended cancer treatment. The investigators will use theory-informed multilevel strategies to create the AYAHIV Role-based Responsibilities for Oncology-focused Workforce (ARROW) program to increase uptake of services for early diagnosis and improve compliance with cancer treatment for KS, NHL, and CC. Our overall approach is based on the evidence-based strategy of peer support for engagement and learning. At the individual level, the investigators will address barriers by embedding peer counselors to support AYAHIV. At the provider level, the investigators will create a peer-to-peer learning network to build linkages between those specializing in pediatric and adult HIV treatment and cancer care. At the health care system level, the investigators will bring together health care administrators and Zambian Ministry of Health policy makers to review barriers and to develop and implement collaborative solutions. The investigators will use implementation science methods to evaluate effectiveness, implementation outcomes, and cost-effectiveness of the ARROW program compared with a one-time education campaign by pursuing the following aims:

Aim 1. Conduct randomized trials to compare the ARROW program with the one-time education campaign in increasing services received by AYAHIV to facilitate early diagnosis (physical exam for KS and NHL, CC screening, and timely diagnostic testing) and in improving adherence to cancer treatment.

Aim 2. Use mixed methods to assess implementation outcomes of the ARROW program compared with one-time education based on acceptability, feasibility, appropriateness, fidelity, and sustainability.

Aim 3. Perform economic evaluations to assess cost-effectiveness and return-on-investment scenarios.

Successful completion of these aims will yield a set of data-driven strategies that can be scaled up to reduce premature cancer mortality among AYAHIV. To support future implementation efforts, the investigators will generate incremental cost-effectiveness estimates, conduct policy simulations, evaluate implementation outcomes, and assess challenges and facilitators to optimize the ARROW program. The model tested in Zambia can serve as a blueprint for other Sub-Saharan African countries to ensure AYAHIV receive optimal services to facilitate early diagnosis and ensure completion of guideline-recommended treatments. The ARROW program will also provide a framework for implementing expanded services, such as preventive services and survivorship care, to further reduce the burden of cancer AYAHIV face.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 39 years of age at the time of study enrolment, on antiretroviral medication (ART) for at least 6 months and with no pending plans to move from current residence during the 3-year study duration

Exclusion Criteria:

* pregnant at study enrolment

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion who complete screening/physical examination | 12 months after study enrollment
  Number who complete screening/physician exams
Proportion who complete recommended cancer treatment modalities | 12 months after diagnosis
  Number who complete treatment

SECONDARY OUTCOMES:
Proportion who complete recommended follow-up supplemental diagnostic procedures | 3 months from receipt of follow-up referral
  Number who complete follow-up
Proportion who initiate cancer treatment | 3 months from diagnosis
  Number who initiate treatment
Proportion alive at 12 months | 12 months after diagnosis
  Number alive at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Facilities, Lusaka, Zambia